CLINICAL TRIAL: NCT01400516
Title: Teriparatide for Joint Erosions in Rheumatoid Arthritis: The TERA Trial
Acronym: TERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Daniel H. Solomon, M.D.,MPH, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010P002691
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Bone erosion; Osteopenia
MeSH Terms: conditions — Arthritis, Rheumatoid; Bone Diseases, Metabolic | interventions — Teriparatide; Calcium Citrate; Vitamin D; Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teriparatide (Experimental): The participants who are in treatment arm received teriparatide 20 μg, subcutaneous injection, 1 injection per day, with a biologic for 12 months. A second year of teriparatide was offered to all interested participants. All participants received daily 1000 milligrams (mg) of calcium citrate, 800 IU of vitamin D and a Tumor Necrosis Factor (TNF) antagonist.
  Interventions: Drug: Teriparatide; Drug: calcium citrate; Drug: Vitamin D; Drug: TNF antagonist
- Control Arm (Other): The participants randomized to the control arm had the same testing as those in the treatment arm and were offered teriparatide, if determined to be effective in healing bone erosions, after the first 12 months. All participants received daily 1000 mg of calcium citrate, 800 IU of vitamin D and a TNF antagonist.
  Interventions: Drug: calcium citrate; Drug: Vitamin D; Drug: TNF antagonist

INTERVENTIONS:
Drug: Teriparatide — 20 μg, subcutaneous injection, 1 injection per day
  Other Names: Forteo
  Arms: Teriparatide
Drug: calcium citrate — 1000 mg of calcium citrate
Drug: Vitamin D — 800 IU of Vitamin D
Drug: TNF antagonist — TNF antagonist as prescribed in clinical practice (such as etanercept or adalimumab)

SUMMARY:
Summary:

The investigators propose a randomized controlled open label study of teriparatide in men or women with rheumatoid arthritis and joint erosions. Specifically, the investigators will examine whether teriparatide in combination with a biologic can retard the development of joint erosions. The study will be conducted at Brigham and Women's Hospital Arthritis Center, several Brigham and Women's Hospital Arthritis Center satellite practices, the University of Massachusetts Medical Center, and Massachusetts General Hospital.

Hypothesis:

The investigators hypothesize that the combination of teriparatide with biologic will be much more effective at retarding erosion progression then a biologic alone.

DETAILED DESCRIPTION:
I. Introduction:

While generalized osteoporosis causes tremendous disability in patients with Rheumatoid Arthritis (RA) and occurs relatively frequently in such patients, there has been little research on treatments for osteoporosis in patients with RA. Not only are there important questions about the effects of teriparatide on Bone Mineral Density (BMD) in patients with RA, but little is known about how it might affect localized bone erosions or RA disease activity.

Recent data in a mouse model of RA suggest that intermittent para-thyroid hormone (PTH) in the setting of potent immunosuppressives may indeed heal bone erosions. This study showed an additive effect of PTH in addition to a biologic on erosion healing. To the best of our knowledge, this has yet to be demonstrated in humans. That is the primary aim of the proposed study.

II. Objectives and Hypotheses:

To assess the effects of teriparatide among a group of patients with RA and erosions, all using biologics, with respect to:

1. Joint erosion volume by 3-dimensional computed tomography (3D CT) scan;
2. Lumbar BMD by dual-energy X-ray absorptiometry (DXA);
3. Hip BMD by DXA; and
4. RA disease activity measured by the Disease Activity Score (DAS) and acute phase reactants.

The hypotheses to be tested include:

1. Joint erosion scores, measured by 3D CT scan, will be significantly improved at study completion in patients taking teriparatide.
2. Teriparatide will significantly increase BMD at all sites as measured by DXA.
3. RA disease activity measures will be stable during the study year.

III. Statistical Analyses:

The total erosion volume will be calculated for each hand/wrist and for each of the six sub-regions: radius, ulna, proximal carpals [scaphoid, lunate, triquetrum, and pisiform), distal carpals (capitate, hamate, trapezium, trapezoid, and the carpometacarpal (CMC) joints), metacarpophalangeal (MCP) joints, and proximal interphalangeal (PIP) joints. We will perform the hand level-analysis with the individual hands as our study units. In a pre-trial study, repositioning reproducibility was excellent at the hand-level (N = 10) as noted in Duryea et al (REF ). The average total erosion volume in a single hand/wrist was 428.1 mm^3. Average erosion volume was smallest at the ulna (6.4 mm^3) and largest in the distal carpals (144.8 mm^3). The intra-class correlation (ICC) values were excellent, ranging from 0.97 to 1.00. The root mean square stand deviation (RMSSD) was 31.2 mm^3 with a coefficient of variation (CoV) of 7.3%. The CoVs for the six measured hand regions ranged from 7.6% to 21.0%. Individual regions with increased erosion volume tended to have correspondingly larger RMSSD values, while the dependence of the CoV on the total volume was less pronounced.

The outcome for the primary analysis will compare the changes in erosion volume from baseline to follow-up for the subjects receiving teriparatide versus those not. If we find that the change in whole hand erosion volume is significantly better for teriparatide users than controls, then we will have met the primary outcome. In a secondary analysis, we will assess the change in erosion volume at each of the six anatomic sites. As these are secondary analyses, no correction for multiple testing will be pursued. Significance at the whole hand and anatomic site level will be based on a two-tail test of significance with a p-value < 0.05 considered statistically significant.

For all analyses, we will analyze the data at the level of the hand, adjusting for within subject correlation between the two hands using a generalized linear mixed model (GLMM). Baseline subject characteristics will be compared between the two groups using two sample t tests, Chi-square tests or non-parametric tests when applicable. Characteristics of interest include age, gender, duration of RA, serologic status [rheumatoid factor (RF) positive and anti-citrullinated protein antibody (ACPA) positive], use of oral corticosteroids, use of concomitant non-biologic disease-modifying antirheumatic drugs (DMARDs), baseline DAS score, baseline Total Sharp Score, and baseline health assessment questionnaire (HAQ) score. If any of these characteristics are found to be imbalanced across groups (p-value < 0.10), those variables will be introduced as possible covariates in the model. However, for this small study with 48 hands, the final model will include no more than 5 predictors.

Several exploratory subgroup analyses will be pursued. These include subgroups of patients based on/with:

* Corticosteroid users or not at baseline;
* Less than or greater than 2 years of RA at baseline;
* In RA remission, defined in three ways: as DAS28 ≤ 2.6, simple disease activity index (SDAI) ≤ 3.3, and boolean [swollen joint count (SJC), tender joint count (TJC), patient global and c-reactive protein (CRP) ≤ 1];
* high sensitivity CRP (hsCRP) < 3mg/L versus ≥ 3mg/L;
* Less than median # of erosions (based on Sharp Score) versus greater than;
* Less than median erosion volume at baseline versus greater than; and
* Depth of erosion: 25% deepest erosions versus other erosions.

The secondary analyses will all be considered exploratory and will follow the same analytic strategy as the primary analyses. Due to small sizes, unadjusted GLMM model will be used in sub-group analyses.

Analyses of secondary outcomes noted above will also be considered exploratory. They will also follow the same analytic strategy as the primary analyses.

If follow up is less than complete, we will estimate the effect under intention-to-treat. Several missing value techniques will be applied to impute the missing outcomes including last observation carried forward, single imputation (e.g. replacing missing values with the sample mean or median), and multiple imputation. Sensitivity analysis will compare these methods with complete case analysis.

IV. Sample Size Estimates:

We have used the estimates derived from the pre-trial replication study to estimate sample size for the trial. We considered analyses both at the level of the subject and at the level of the individual hand. Assessing individual hands provides twice as many observations (two hands for each patient), but these observations are not independent of one another. In our pilot analysis that evaluated 5 patients (10 hands), log-transformation was applied to total volumes to achieve an approximately normal distribution. The average value of log-transformed total volume was 5.32, with standard deviation of 1.34. Assuming that a reasonable ICC between two hands/wrists, on the same patient ranges from 0.20 to 0.50, we estimated the sample size required to achieve 80% power, given a range of differences with a significance level of 0.050 using a two-sided test (see Table 2) 17. To detect a moderate difference of 15%-25% between groups, the sample size needed to achieve adequate statistical power would range from 10 to 34 per study group.

We recruited 12 patients per group (24 hands), assuming an ICC of 0.5.

ELIGIBILITY:
Inclusion Criteria:

All men and women 45 years of age or older with RA and joint erosions by plain x-ray who are taking a biologic for at least three months and who have not taken more than two weeks of a bone active agent in the last 12 months will be eligible and screened for their interest in participating in the proposed randomized trial.

1. RA will be defined according to the 2010 American College of Rheumatology/European League Against Rheumatism diagnostic and classification criteria.
2. Osteopenic bone mineral density will be defined as a t-score between -1.0 and -2.5 on either a DXA of the posteroanterior (PA) or lateral lumbar spine or the femoral neck or total hip. Potential subjects with prior minimal trauma fractures will be excluded.

   2.Subjects must be able to give written informed consent.

Exclusion Criteria:

1. A switch in DMARD in the last 3 months;
2. Current use of chronic oral glucocorticoids > 5 milligrams per day;
3. A prior history of intolerance to teriparatide;
4. T-score < -2.5 or a prior minimal trauma fracture;
5. Use of a bone active agent for over 2 weeks in the last 12 months (these agents include oral and intravenous bisphosphonates, hormone replacement therapy, calcitonin, raloxifene, teriparatide, suppressive doses of thyroxine, lithium, pharmacological doses of vitamin D (greater than 2000 IU/day or anticonvulsants);
6. History of significant cardiac, hepatic, current alcohol abuse, or major psychiatric disorders;
7. Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including hematologic malignancies and solid tumors, except basal cell carcinoma of the skin that has been excised and cured), or breast cancer diagnosed within the previous 20 years;
8. No current diagnoses of disorders known to affect bone metabolism including hyperthyroidism, hyperparathyroidism, osteomalacia, or Paget's disease. All participants will be required to have normal serum levels of 25-OH vitamin D (> 20 ng/ml), intact PTH, and thyroid stimulating hormone (TSH). If PTH and/or 25-hydroxy vitamin D (25-OH D) levels are abnormal, subjects may be given calcium and/or multivitamin supplements and be re-tested in 2-12 weeks;
9. Serum calcium (Ca) > 10.6 mg/dl,and 24-hour urine calcium > 400 mg. If minor abnormalities are detected in any of these parameters, the test may be repeated;
10. Patients who have had external beam radiation; and
11. Patients currently on digoxin.
12. Women that are currently pregnant or breast-feeding or plan on becoming pregnant over the course of participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2015-07-30 (Actual); Study Completion 2016-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Solomon, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Ellen M. Gravallese, MD, Principal Investigator — University of Massachusetts, Worcester; Jonathan Kay, MD, Principal Investigator — University of Massachusetts, Worcester; Marcy B. Bolster, M.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts

REFERENCES:
- [Background] Rasch EK, Hirsch R, Paulose-Ram R, Hochberg MC. Prevalence of rheumatoid arthritis in persons 60 years of age and older in the United States: effect of different methods of case classification. Arthritis Rheum. 2003 Apr;48(4):917-26. doi: 10.1002/art.10897. PMID 12687533
- [Background] Haugeberg G, Uhlig T, Falch JA, Halse JI, Kvien TK. Bone mineral density and frequency of osteoporosis in female patients with rheumatoid arthritis: results from 394 patients in the Oslo County Rheumatoid Arthritis register. Arthritis Rheum. 2000 Mar;43(3):522-30. doi: 10.1002/1529-0131(200003)43:33.0.CO;2-Y. PMID 10728744
- [Background] Hooyman JR, Melton LJ 3rd, Nelson AM, O'Fallon WM, Riggs BL. Fractures after rheumatoid arthritis. A population-based study. Arthritis Rheum. 1984 Dec;27(12):1353-61. doi: 10.1002/art.1780271205. PMID 6508860
- [Background] Michel BA, Bloch DA, Wolfe F, Fries JF. Fractures in rheumatoid arthritis: an evaluation of associated risk factors. J Rheumatol. 1993 Oct;20(10):1666-9. PMID 8295176
- [Background] Spector TD, Hall GM, McCloskey EV, Kanis JA. Risk of vertebral fracture in women with rheumatoid arthritis. BMJ. 1993 Feb 27;306(6877):558. doi: 10.1136/bmj.306.6877.558. No abstract available. PMID 8461772
- [Background] Hall GM, Spector TD, Griffin AJ, Jawad AS, Hall ML, Doyle DV. The effect of rheumatoid arthritis and steroid therapy on bone density in postmenopausal women. Arthritis Rheum. 1993 Nov;36(11):1510-6. doi: 10.1002/art.1780361105. PMID 8240428
- [Background] Cooper C, Coupland C, Mitchell M. Rheumatoid arthritis, corticosteroid therapy and hip fracture. Ann Rheum Dis. 1995 Jan;54(1):49-52. doi: 10.1136/ard.54.1.49. PMID 7880122
- [Background] Saag KG, Emkey R, Schnitzer TJ, Brown JP, Hawkins F, Goemaere S, Thamsborg G, Liberman UA, Delmas PD, Malice MP, Czachur M, Daifotis AG. Alendronate for the prevention and treatment of glucocorticoid-induced osteoporosis. Glucocorticoid-Induced Osteoporosis Intervention Study Group. N Engl J Med. 1998 Jul 30;339(5):292-9. doi: 10.1056/NEJM199807303390502. PMID 9682041
- [Background] Cohen S, Levy RM, Keller M, Boling E, Emkey RD, Greenwald M, Zizic TM, Wallach S, Sewell KL, Lukert BP, Axelrod DW, Chines AA. Risedronate therapy prevents corticosteroid-induced bone loss: a twelve-month, multicenter, randomized, double-blind, placebo-controlled, parallel-group study. Arthritis Rheum. 1999 Nov;42(11):2309-18. doi: 10.1002/1529-0131(199911)42:113.0.CO;2-K. PMID 10555025
- [Background] Adachi JD, Bensen WG, Brown J, Hanley D, Hodsman A, Josse R, Kendler DL, Lentle B, Olszynski W, Ste-Marie LG, Tenenhouse A, Chines AA. Intermittent etidronate therapy to prevent corticosteroid-induced osteoporosis. N Engl J Med. 1997 Aug 7;337(6):382-7. doi: 10.1056/NEJM199708073370603. PMID 9241127
- [Background] Lane NE, Sanchez S, Modin GW, Genant HK, Pierini E, Arnaud CD. Parathyroid hormone treatment can reverse corticosteroid-induced osteoporosis. Results of a randomized controlled clinical trial. J Clin Invest. 1998 Oct 15;102(8):1627-33. doi: 10.1172/JCI3914. PMID 9788977
- [Background] Eggelmeijer F, Papapoulos SE, van Paassen HC, Dijkmans BA, Valkema R, Westedt ML, Landman JO, Pauwels EK, Breedveld FC. Increased bone mass with pamidronate treatment in rheumatoid arthritis. Results of a three-year randomized, double-blind trial. Arthritis Rheum. 1996 Mar;39(3):396-402. doi: 10.1002/art.1780390307. PMID 8607888
- [Derived] Solomon DH, Kay J, Duryea J, Lu B, Bolster MB, Yood RA, Han R, Ball S, Coleman C, Lo E, Wohlfahrt A, Sury M, Yin M, Yu Z, Zak A, Gravallese EM. Effects of Teriparatide on Joint Erosions in Rheumatoid Arthritis: A Randomized Controlled Trial. Arthritis Rheumatol. 2017 Sep;69(9):1741-1750. doi: 10.1002/art.40156. Epub 2017 Jul 14. PMID 28544807
- See also: Brigham and Women's Clinical Trials — http://www.brighamandwomens.org/research/clinical/volunteer.aspx

RESULTS

PARTICIPANT FLOW:
Period: Primary Trial
Arm/Group | Control Arm | Teriparatide
Started | 12 | 14
Completed | 12 | 12
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Extension Trial
Arm/Group | Control Arm | Teriparatide
Started | 6 (Only 6 participants in the Control arm entered the Extension Trial.) | 7 (Only 7 participants in the Teriparatide arm entered the Extension Trial.)
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis includes 24 participants who were randomized, 2 participants withdrew prematurely and are not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Teriparatide | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [56 to 65] | 63 [56 to 69] | 62 [56 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Joint Erosion Volume Measured by 3-Dimensional Computed Tomography (3D CT) Scan
Description: Both hands were scanned using a CT scanner. A semi-automated software tool was used to segment the erosion margins in 3D. A board certified radiologist identified the individual erosions in six sub-regions: radius, ulna, proximal carpals, distal carpals, metacarpophalangeal (MCP) joints and proximal interphalangeal (PIP) joints. The average total in a single hand/wrist was calculated. A negative change from Baseline(less joint erosions) indicates improvement.
Time Frame: Baseline and Month 12
Population: Analysis includes 24 participants who were randomized, 2 participants withdrew prematurely and are not included.
Measure: Median (Inter-Quartile Range); unit: cubic millimeter (mm^3)
Arm/Group | Control Arm | Teriparatide
Number analyzed (Participants) | 12 | 12
cubic millimeter (mm^3)
  Baseline | 571.4 [160.0 to 1341.6] | 369.8 [171.0 to 1163.9]
  Change from Baseline at Month 12 | 9.1 [-29.6 to 26.4] | -0.4 [-34.5 to 29.6]
Statistical Analysis 1: Comparison: Control Arm vs Teriparatide; Test type: Superiority; p = 0.28, Linear mixed model — A p-value < 0.05 is considered statistically significant; Median Difference (Final Values) = 9.5 — control-teriparatide

2. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) Measured by Dual-Energy X-ray Absorptiometry (DXA) and Instant Vertebral Assessment (IVA) Scan
Description: BMD was measured at the lumbosacral spine antero-posterior and at the femoral neck using a densitometer. A positive change from Baseline (increased bone density) indicates improvement.
Time Frame: Baseline and Month 12
Population: Analysis includes 24 participants who were randomized, 2 participants withdrew prematurely and are not included.
Measure: Mean (Standard Deviation); unit: grams/centimeters squared (g/cm^2)
Arm/Group | Control Arm | Teriparatide
Number analyzed (Participants) | 12 | 12
grams/centimeters squared (g/cm^2)
  Spine, Baseline | 0.93 (0.11) | 0.91 (0.09)
  Spine, Change from Baseline at Month12 | -0.002 (0.11) | 0.06 (0.04)
  Femoral neck, Baseline | 0.73 (0.09) | 0.68 (0.06)
  Femoral neck, Change from Baseline at Month 12 | -0.03 (0.08) | 0.03 (0.03)

3. Secondary Outcome: Change From Baseline in Disease Activity Score 28 Joint Count C-Reactive Protein (DAS-28 CRP)
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and C-Reactive Protein (CRP) for a total possible score of 2 to 10. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline and Month 12
Population: Analysis includes 24 participants who were randomized, 2 participants withdrew prematurely and are not included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Teriparatide
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 2.73 (1.19) | 2.66 (1.43)
  Change from Baseline at Month 12 | -0.50 (0.67) | 0.42 (0.67)

ADVERSE EVENTS:
Time Frame: Up to 2 Years
Description: Analysis includes 24 participants who were randomized, 2 participants withdrew prematurely and are not included.
Arm/Group | Control Arm | Teriparatide
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 2/12 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=12) | Teriparatide (N=12)
Death (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control Arm (N=12) | Teriparatide (N=12)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hair lost (Skin and subcutaneous tissue disorders) | 0 | 2
High serum calcium (Investigations) | 0 | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Pain in knees and ankles (Musculoskeletal and connective tissue disorders) | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes